CLINICAL TRIAL: NCT06476106
Title: Mitigating Headward Fluid Shifts With Venoconstrictive Thigh Cuffs During Spaceflight
Brief Title: Human Research Program Flight Thigh Cuff
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000453
Record Dates: First submitted 2024-03-07; First posted 2024-06-26 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flight Thigh Cuff Crew Participants (Experimental): Participants will participate in 2 preflight study sessions consisting of a VTC fit check and a baseline data collection without and with the VTC donned. Participants will also participate in 3 inflight study sessions: a VTC fit check on flight day 30 (FD30) and two separate data collection sessions on flight day 45 (FD45) and 45 days before landing (R-45). During the two in-flight data collection days, participants will be studied before and for up to 6 hours after donning the VTC.
  Interventions: Device: Venoconstrictive Thigh Cuff (VTC)

INTERVENTIONS:
Device: Venoconstrictive Thigh Cuff (VTC) — The VTC is an adjustable fabric cuff that is worn on the upper thighs to retain some fluid in the legs. It consists of wide straps and a buckle which allow it to be tightened, then velcro to secure the strap in the tightened position. There is also lacing that can be tightened for micro adjustments. Imbedded within the fabric strap is a bladder that is not used for increasing tightness but allows the pressure of the cuff to be measured and tracked.
  Other Names: Thigh Cuff

SUMMARY:
Venoconstrictive Thigh Cuffs (VTC) are being evaluated to determine the effectiveness at reversing the headward fluid shift that occurs during weightlessness. If successful, future studies may be done to implement these as a CM to SANS. To support this effort, participants will participate in 2 preflight study sessions consisting of a VTC fit check and a baseline data collection without and with the VTC donned. Participants will also participate in 3 inflight study sessions: a VTC fit check on flight day 30 (FD30) and two separate data collection sessions on flight day 45 (FD45) and 45 days before landing (R-45). During the two in-flight data collection days, participants will be studied before and for up to 6 hours after donning the VTC.

ELIGIBILITY:
Inclusion Criteria:

* Astronauts participating in missions that are ≥2 months

Exclusion Criteria:

* Having known allergies to proparacaine hydrochloride ophthalmic solution precludes participation in this study
* Use of ethinyl estradiol Combined Oral Contraceptive (COC) pills precludes participation in this study
* Having increased risk of venothromboembolism (VTE) based on preflight thrombosis/clotting related biomarkers precludes participation in this study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2028-05-14 (Estimated); Study Completion 2030-05-14 (Estimated)

PRIMARY OUTCOMES:
Internal Jugular Vein (IJV) area | Thigh Cuff Measures 90 days before mission, after 45 days in mission, and 45 days before return
  Measured using Ultrasound.
IJV pressure | Thigh Cuff Measures 90 days before mission, after 45 days in mission, and 45 days before return
  Measured using the VeinPres device during Ultrasound.
Intraocular Pressure (IOP) | Thigh Cuff Measures 90 days before mission, after 45 days in mission, and 45 days before return
  Measured using the Pneumatonometer.
stroke volume | Thigh Cuff Measures 90 days before mission, after 45 days in mission, and 45 days before return
  Measured from data collected during Ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon R Macias, PhD, Principal Investigator — National Aeronautics and Space Administration (NASA)
Locations (1):
- Johnson Space Center, National Aeronautics and Space Administration, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No